CLINICAL TRIAL: NCT06598293
Title: Routine Electronic Patient-reported Outcome Measures During and After Radiotherapy: A Randomized Controlled Study (REPROM)
Brief Title: Routine Electronic Patient-reported Outcome Measures During and After Radiotherapy: A Randomized Controlled Study
Acronym: REPROM
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hwa Kyung Byun, Professor, Yonsei University
Other Study IDs: 9-2024-0095
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group: REPROM group: Subjects in the test group will self-report symptoms that occur using smartphones before radiotherapy, once a week during treatment, at the end of treatment, once a week until one month after treatment, and at 1 month and 3~6 months after treatment (PRO-CTCAE, Pain NRS). The radiation oncologist will identify the symptoms reported in the REPROM and take appropriate medical measures to improve the symptoms based on this.
  A survey alert will be sent to the patient at the time of REPROM implementation, and the subject will self-report the patient's symptoms through the mobile messenger KakaoTalk using a smartphone. The survey data is automatically sent to the EMR and can be checked by the attending physician at the time of consultation. A score of 4 or higher will be automatically alerted to the attending physician and the research nurse, and the research nurse may contact the subject if necessary and recommend additional care to the attending physician.
  Interventions: Behavioral: PRO-CTCAE, Pain NRS
- Control group: Standard care group: Control subjects receive standard care without self-report of REPROM. Both groups may receive appropriate medical attention for the symptoms observed at the time of examination.
  Both groups will administer HR-QOL questionnaires (EORTC-QLQ-C30, EQ-5D-5L, EQ-VAS) before radiotherapy, at the end of treatment, 1 month after treatment, and 3~6 months after treatment.

INTERVENTIONS:
Behavioral: PRO-CTCAE, Pain NRS — The Common Terminology Criteria for Adverse Events (PRO-CTCAE) is a PROM developed to systematically and objectively reflect patients' experiences and perceptions of therapeutic drugs in toxicity evaluation and adverse event reporting. PRO-CTCAE can be used to monitor patients' symptoms and side effects, support therapeutic decision-making, facilitate communication among medical staff, implement patient-centred care, and screen for health conditions.
  Groups: Test group: REPROM group

SUMMARY:
Patients in this study will be asked to periodically self-report their symptoms using their smartphones during the radiotherapy period and during the acute phase (3 months) after treatment, and radiation oncology physicians will evaluate the impact on cancer patients' quality of life and determine whether they can improve health outcomes by using this data in their practice.

DETAILED DESCRIPTION:
The purpose of this study is to determine the efficacy, feasibility, and acceptability of routine PROM reporting using smartphones during treatment and during the acute phase after treatment in patients undergoing radiotherapy.

Subjects who voluntarily consent to the study will be assigned to either the test group or the control group through randomization.

• Test group: REPROM group Subjects in the test group will self-report symptoms that occur using smartphones before radiotherapy, once a week during treatment, at the end of treatment, once a week until one month after treatment, and at 1 month and 3~6 months after treatment (PRO-CTCAE, Pain NRS). The radiation oncologist will identify the symptoms reported in the REPROM and take appropriate medical measures to improve the symptoms based on this.

A survey alert is sent to the patient at the time of REPROM implementation, and the subject uses a smartphone to conduct a self-report questionnaire on patient symptoms sent through the mobile messenger KakaoTalk as shown in the screenshot below. The survey data is automatically sent to the EMR and can be checked by the attending physician at the time of consultation. A score of 4 or higher will be automatically alerted to the attending physician and the research nurse, and the research nurse may contact the subject if necessary and recommend additional care to the attending physician.

• Control group: Usual care group Control subjects receive usual care without self-report of REPROM. Subjects in both groups may receive appropriate medical attention for the symptoms observed at the time of treatment. Subjects in both groups will be asked to take HR-QOL questionnaires (EORTC-QLQ-C30, EQ-5D-5L, EQ-VAS) before radiotherapy, at the end of treatment, at 1 month after treatment, and at 3~6 months after treatment.

*Study design: a prospective randomized parallel-group pilot study

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Histologically confirmed diagnosis of cancer
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* The ability to own and use a smartphone

Exclusion Criteria:

* Terminal cancer
* Cognitive impairment
* Not using your smartphone

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean patients who visited the hospital and will receive treatment from the radiation oncology department
Sampling Method: Non-Probability Sample
Enrollment: 536 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean change score from baseline in Quality of Life Assessment Tool (EORTC-QLQ-C30) | 36 months after registration
  Comparison of quality of life assessment tool scores between groups is performed using independent t-test. Linear mixed-effect model is used in the intention-to-treat study population. Age, sex, pretreatment PROM score, cancer type, and stage are controlled as fixed covariates, and radiation oncology and attending physician are controlled as random intercepts. For sensitivity analysis, additional analysis is performed on patients who completed more than 80% of the REPROM questionnaire. Since this study is an exploratory analysis, a two-sided significance level of .05 is used for all comparisons without redundancy adjustment.

CONTACTS AND LOCATIONS:
Overall Officials: Hwakyung BYUN, Phd, Principal Investigator — Severance Hospital
Locations (1):
- Yongin Severance Hospital, Yongin-si, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holch P, Absolom KL, Henry AM, Walker K, Gibson A, Hudson E, Rogers Z, Holmes M, Peacock R, Pini S, Gilbert A, Davidson S, Routledge J, Murphy A, Franks K, Hulme C, Hewison J, Morris C, McParland L, Brown J, Velikova G. Online Symptom Monitoring During Pelvic Radiation Therapy: Randomized Pilot Trial of the eRAPID Intervention. Int J Radiat Oncol Biol Phys. 2023 Mar 1;115(3):664-676. doi: 10.1016/j.ijrobp.2022.09.078. Epub 2022 Oct 12. PMID 36241128
- [Background] Bae WK, Kwon J, Lee HW, Lee SC, Song EK, Shim H, Ryu KH, Song J, Seo S, Yang Y, Park JH, Lee KH, Han HS. Feasibility and accessibility of electronic patient-reported outcome measures using a smartphone during routine chemotherapy: a pilot study. Support Care Cancer. 2018 Nov;26(11):3721-3728. doi: 10.1007/s00520-018-4232-z. Epub 2018 May 7. PMID 29732483
- [Result] Steinbeck V, Langenberger B, Schoner L, Wittich L, Klauser W, Mayer M, Kuklinski D, Vogel J, Geissler A, Pross C, Busse R. Electronic Patient-Reported Outcome Monitoring to Improve Quality of Life After Joint Replacement: Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Sep 5;6(9):e2331301. doi: 10.1001/jamanetworkopen.2023.31301. PMID 37656459